CLINICAL TRIAL: NCT04589195
Title: Measurement of an Application - Based Delivery of Mindfulness Training Program Content
Brief Title: Measuring Mindfulness Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Amishi Jha, Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20201140
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Cognitive Change
Keywords: Mindfulness Training; Cognitive Training; Psychological Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Training (MT) Group (Experimental): Participants will receive four weeks of MT.
  Interventions: Behavioral: Mindfulness Training
- Wait List MT Group (Active Comparator): Participants will receive four weeks of MT training after a five week washout period.
  Interventions: Behavioral: Mindfulness Training

INTERVENTIONS:
Behavioral: Mindfulness Training — The intervention includes four weeks of MT application use, accessed via phone or computer, consisting of 15-minute daily mindfulness practices 5 days a week.

SUMMARY:
The purpose of the research study is to learn more about how ROTC cadets may engage with mindfulness training program content that is delivered through a smartphone or website application. Mindfulness training program content includes mindfulness practices that foster attention and awareness.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are between 18 and 64 years of age.
2. Individuals who are fluent English speakers.
3. Individuals who have access to either an Apple or Android smart phone and a desktop or laptop computer, are able to adequately and independently use both devices, and have Internet connection.
4. Individuals who are willing and able to consent to participate in the study.
5. Individuals who are in the South Florida ROTC program.

Exclusion Criteria:

1.Individuals with an active and untreated mental condition (e.g., Bipolar disorder, Major Depression) and/or hospitalization for psychological/mental health issues within the last month.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-12-26 (Actual)

PRIMARY OUTCOMES:
Change in Positive Affect | Baseline to Week 5
  Positive affect will be measured with the 10-item version of the Positive and Negative Affect Schedule (PANAS-10). The PANAS positive sub-scale has 5 items and a range of scores from 5 to 25, with a higher score indicating a higher positive mood.
Change in Negative Affect | Baseline to Week 5
  Negative affect will be measured with the 10-item version of the Positive and Negative Affect Schedule (PANAS-10). The PANAS negative sub-scale has 5 items and a range of scores from 5 to 25, with a higher score indicating a higher negative mood.
Change in Perceived Stress | Baseline to Week 5
  Perceived Stress will be measured with the Perceived Stress Scale (PSS). PSS has a range of scores from 0 to 40, with a higher score indicates a higher level of perceived stress.

SECONDARY OUTCOMES:
Change in Sustained Attention Response Task (SART) scores | Baseline to Week 5
  The SART involves pressing a button to frequently presented non-target trials and withholding the button press to the infrequent target trials. The participants can have a total score between 0 and 100%, with a higher score indicating butter sustained attention.
Change in Cognitive Failures | Baseline to Week 5
  Cognitive Failures will be measured with the Cognitive Failures Questionnaire (CFQ). CFQ has a range of scores from 0 to 100, with a higher score indicating more cognitive failures.

OTHER OUTCOMES:
Change in Psychological Health | Baseline to Week 5
  Patient Health Questionnaire (PHQ4) will be used to assess depression and anxiety. PHQ has a range of scores from 0 to 12, with a higher score indicating higher level of depression and anxiety.
Change in Mindfulness | Baseline to Week 5
  Mindfulness will be measured with the short 15-item version of the Five-Facet Mindfulness Questionnaire (FFMQ-15). FFMQ-15 has a range of scores from 15 to 75, with a higher score indicating a greater level of mindfulness.
Change in Decentering | Baseline to Week 5
  Decentering will be measured with the decentering scale from the Experience Questionnaire (EQ-D). EQ-D has a range of scores from 11 to 55, with a higher score indicating a greater level of decentering.

CONTACTS AND LOCATIONS:
Overall Officials: Amishi Jha, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No